CLINICAL TRIAL: NCT05968638
Title: Single-Blind Randomized Ketogenic Diet vs. Control Diet in People With Schizophrenia
Brief Title: Ketogenic Diet in People With Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Chief and Director, Treatment Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00106193
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Diet; Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive either a ketogenic diet or regular diet
Who Masked: Investigator, Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Diet (Placebo Comparator)
  Interventions: Other: Regular Diet
- Ketogenic Diet (Active Comparator)
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Regular Diet — Regular Diet
  Arms: Regular Diet
Other: Ketogenic Diet — Ketogenic Diet
  Arms: Ketogenic Diet

SUMMARY:
Schizophrenia is a serious mental disorder with a heterogenous presentation, lack of clear understanding of pathophysiology and only partially effective treatments. First-line antipsychotic drugs block dopamine, but many people continue to suffer from persistent positive or negative symptoms that cannot be fully treated with available medications. Recently, our group has found that dietary modulations have efficacy comparable to antipsychotic medications and that determining which patients could benefit from a personalized treatment framework is critical.

The ketogenic diet consists of low-carbohydrate, moderate protein and high fat intake inducing a state in which ketone bodies in the blood provide energy to the cells. In pharmacologic mouse models a ketogenic diet regimen resulted in complete restoration of normal behaviors, independent of strict caloric restriction and other work has suggested that a ketogenic diet may improve schizophrenia like deficits in rodents. An open label ketogenic diet study in the 1950s reported improvement in schizophrenia symptom. At least 7 additional case reports have found robust improvements or complete resolution of schizophrenia symptoms. Recently a retrospective study found robust and significant improvements in schizophrenia symptoms in 10 schizoaffective disorder patients treated with a ketogenic diet. In addition to psychiatric symptoms, improvements in metabolic outcomes have been demonstrated. However, to date, there have been no published double blind randomized controlled trials evaluating the effects of a ketogenic diet since few sites can conduct inpatient trials and have observation and control for food intake

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 64 years
2. Diagnostic and Statistical Manual (DSM-IV/DSM 5) diagnosis of schizophrenia or schizoaffective disorder
3. Antipsychotic regimen with no dose change in last 14 days
4. Minimum score of 45 on BPRS
5. Body mass index > 18.5
6. Ability to consent determined by a score of 10 or greater on the Evaluation to Sign Consent.

Exclusion Criteria:

1. Pregnant or lactating females
2. Type I diabetes or insulin dependent Type II diabetes
3. Current diagnosis of DSM 5 eating disorder
4. Heart failure
5. corrected QT interval (QTc) prolongation greater than or equal to 500ms
6. Significant kidney disease

   Indicators for possible acute kidney injury (AKI) or moderate chronic kidney disease (CKD) based on some factors below. Each is not used individually but a clinician will determine based on the following:
   * Creatinine > 1.3mg/dL
   * Glomerular Filtration Rate (GFR) < 60 mL/min/1.73 m2
   * Renal tubular disorders
   * History of kidney transplantation
7. Significant liver disease.

   Indicators for possible acute or chronic liver disease. Each is not used individually but a clinician will determine based on the following:
   * Prolonged International Normalized Ratio (INR) greater than or equal to 1.5, elevated bilirubin and aminotransferases (3x normal upper limit) and/or Complete Blood Count (CBC) abnormalities (thrombocytopenia, anemia)
   * Physical examination abnormalities (jaundice, icteric sclera, asterixis)
   * Alcohol use disorder (AUD) based on DSM 5 criteria for moderate AUD
   * History of liver disease (cirrhosis, Wilson disease, Gilbert disease, chronic hepatitis, autoimmune hepatitis, primary biliary cirrhosis (PBC), primary Sclerosing Cholangitis (PSC) alpha-1 antitrypsin deficiency, hereditary hemochromatosis, Budd-Chiari syndrome)
   * History of liver transplantation
8. Porphyria
9. Genetic disorders that affect fat metabolism (Gaucher disease, Tay-Sachs disease, medium-chain acyl-CoA dehydrogenase deficiency (MCADD)
10. Carnitine deficiency syndromes (primary carnitine deficiency, carnitine palmitoyltransferase deficiency, carnitine translocase deficiency)
11. Pyruvate kinase deficiency
12. Gastroparesis
13. Refusal to eat intervention diet, food allergies or restrictions that the kitchen cannot accommodate, and/or dietary noncompliance with dietary energy needs

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of positive and negative symptoms | 3 months
  Brief Psychiatric Rating Scale (BPRS): The BPRS scale will be the primary outcome measure. It will be administered at baseline and at the end of each week. The BPRS is considered the most widely used symptom rating scale in psychiatric research, is highly sensitive to change, and has excellent interrater reliability with appropriate training of raters. The BPRS assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe). The score ranges from 18-126, with the higher the number the worse the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D., BCPP, Principal Investigator — Study Principal Investigator
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP), Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No